CLINICAL TRIAL: NCT01279291
Title: Phase 1 Study of Anti-HB-EGF Monoclonal Antibody KHK2866 as Monotherapy in Subjects With Advanced Solid Tumors and in Combination With Chemotherapy in Ovarian Cancer
Brief Title: Study of Anti-HB-EGF Antibody KHK2866 in Subjects With Advanced Solid Tumors and Ovarian Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was stopped due to the inability to determine an acceptable dose with the potential for further study
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Kyowa Hakko Kirin Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2866-US-001
Record Dates: First submitted 2011-01-11; First posted 2011-01-19 (Estimated); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Neoplasms; Ovarian Neoplasms; Fallopian Tube Neoplasms; Primary Peritoneal Neoplasm
Keywords: advanced solid tumor; Ovarian cancer; Primary peritoneal cancer; Fallopian tube cancer
MeSH Terms: conditions — Neoplasms; Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Gemcitabine; Carboplatin; Paclitaxel; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- KHK2866 as monotherapy (Experimental): Groups of subjects will receive a weekly infusions of KHK2866 as treatment for advanced cancer. If there no severe side effects, the dose will be increased for future subjects. A total of four groups are anticipated. Once an acceptable dose is determined an additional seven subjects will be treated at that dose.
  Interventions: Biological: KHK2866
- KHK2866, gemcitabine+carboplatin (Experimental): Open to subjects with ovarian, fallopian tube, or primary peritoneal cancer only.
  One group of subjects will receive one dose below the maximum tolerated dose of KHK2866 identified in Phase 1a along with gemcitabine and carboplatin. The dose of KHK2866 will be increased to the MTD for the next group if no severe side effects are noted. Once an acceptable dose is determined an additional seven subjects will be treated at that dose.
  Interventions: Biological: KHK2866; Drug: Gemcitabine and Carboplatin
- KHK2866, weekly paclitaxel (Experimental): Open to subjects with ovarian, fallopian tube, or primary peritoneal cancer only.
  One group of subjects will receive one dose below the maximum tolerated dose of KHK2866 identified in Phase 1a along with weekly paclitaxel (80 mg/m2). The dose of KHK2866 will be increased to the MTD for the next group if no severe side effects are noted. Once an acceptable dose is determined an additional seven subjects will be treated at that dose.
  Interventions: Biological: KHK2866; Drug: paclitaxel
- KHK2866, pegylated liposomal doxorubicin (Experimental): Open to subjects with ovarian, fallopian tube, or primary peritoneal cancer only.
  One group of subjects will receive one dose below the maximum tolerated dose of KHK2866 identified in Phase 1a along with monthly PLD (40 mg/m2). The dose of KHK2866 will be increased to the MTD for the next group if no severe side effects are noted. Once an acceptable dose is determined an additional seven subjects will be treated at that dose.
  Interventions: Biological: KHK2866; Drug: pegylated liposomal doxorubicin

INTERVENTIONS:
Biological: KHK2866 — Potentially therapeutic monoclonal antibody for the treatment of advanced cancer and ovarian cancer.
Drug: Gemcitabine and Carboplatin — Combination chemotherapy with KHK2866 to treat advanced platinum-sensitive ovarian cancer. Gemcitabine dose 1000 mg/m2, Carboplatin dose AUC=4
  Other Names: Gemzar, Paraplatin
  Arms: KHK2866, gemcitabine+carboplatin
Drug: paclitaxel — Combination chemotherapy with KHK2866 to treat advanced platinum-resistant ovarian cancer. Paclitaxel will be administered weekly at a dose of 80 mg/m2.
  Other Names: Taxol
  Arms: KHK2866, weekly paclitaxel
Drug: pegylated liposomal doxorubicin — Combination chemotherapy with KHK2866 to treat advanced platinum-resistant ovarian cancer. PLD will be administered weekly at a dose of 40 mg/m2.
  Other Names: Doxil
  Arms: KHK2866, pegylated liposomal doxorubicin

SUMMARY:
This is a two-part, Phase 1, open-label, multicenter, dose escalation study of KHK2866 as monotherapy in patients with advanced solid tumors, and in combination with chemotherapy in subjects platinum-sensitive and platinum-resistant ovarian cancer.

DETAILED DESCRIPTION:
During Phase 1a, groups of eligible patients with advanced solid tumors will receive KHK2866 as monotherapy in escalating doses. The Phase 1b portion will enroll patients with ovarian cancer who will receive KHK2866 in combination with one of three chemotherapy regimens (Arms): gemcitabine+carboplatin (platinum-sensitive, weekly paclitaxel (platinum-resistant), or pegylated liposomal doxorubicin (platinum-resistant). Escalating doses of the combination of KHK2866 and the chemotherapy regimen will given to two groups of subjects per Arm. The goal of the study is to learn about the side effects of KHK2866 alone or given in combination with chemotherapy. All subjects will receive study therapy for up to 6 cycles (up to 12 cycles for subjects assigned to PLD [Arm 3 of Phase 1b]), or until disease progression, the development of severe side effects, noncompliance or withdrawal of consent by the subject, or other removal criteria whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented, measurable or non-measurable, advanced primary or recurrent solid tumor (Phase 1a only) which is unresponsive to standard therapy or for which there is no standard therapy available.
* Histologically or cytologically documented ovarian, primary peritoneal, or fallopian tube cancer.
* The subject has objective radiographic disease progression and either unmeasurable or measurable disease during or following the last treatment regimen, or serum cancer antigen-125 (CA-125) greater than 2X the upper limit of normal ([ULN] >70 U/mL
* Life expectancy >3 months.
* Performance status < 3 at study entry.
* Age > 18 years.
* Normal left ventricular ejection fraction.
* Recovered from the effects of recent surgery, radiotherapy, chemotherapy, hormonal therapy, or other therapies for cancer
* Preserved hepatic, renal, and hematopoetic organ function.
* Male and female subjects must use medically accepted contraception.

Exclusion Criteria:

* Ovarian malignancy of low malignant potential.
* Received anti-cancer chemotherapy, hormonal therapy, radiotherapy, immunotherapy, or investigational agents within 4 weeks prior to the first dose of KHK2866 (6 weeks for nitrosourea or mitomycin chemotherapy).
* received Mabs or had major surgery within 4 weeks of the first dose of KHK2866.
* Requires administration of a prohibited medication or treatment including: prophylactic use of erythroid and/or granulocyte colony stimulating factors; concurrent anti-cancer treatment; biologic response modifiers for any condition
* Brain metastases, leptomeningeal or primary brain neoplasm, even if treated.
* Previously untreated or uncontrolled epidural metastasis
* Cerebrovascular accident, Transient ischemic attack; symptomatic head trauma, or seizures or any kind within 6 months
* Dementia, or other disorders of mentation or difficulty speaking or difficulty with comprehension.
* Suspected impending bowel obstruction
* The subject is pregnant,or is lactating.
* Significant uncontrolled intercurrent illness
* Known HIV infection or AIDS-related illness.
* Known active hepatitis B or C or other active liver disease.
* Psychiatric illness, disability or social situation that would compromise the subject's safety, ability to provide consent, or limit his/her compliance with study requirements.
* Experienced a unmanageable hypersensitivity reactions to Mabs or other therapeutic proteins.
* History of second primary cancer, with the exception of: a) curatively resected non-melanomatous skin cancer; b) curatively treated cervical carcinoma in-situ; or c) other primary solid tumor treated with curative intent and no known active disease present and no treatment administered during the last 2 years.
* Additional exclusion criteria for subjects proposed for enrollment into the Phase 1b portion:

  * History of hypersensitivity or infusion reaction to any of the proposed chemotherapy arm's agents that could not be controlled with pre-medication and/or infusion rate adjustment;
  * Prior treatment with KHK2866;
  * History of Grade ≥ 3 non-hematologic or Grade 4 hematologic toxicity attributable to any of the proposed chemotherapy arm's agents
  * For subjects proposed to receive treatment with KHK2866 plus PLD: prior total cumulative exposure to doxorubicin must be ≤ 240 mg/m2.
* Subjects with a known history of interstitial lung disease or pulmonary fibrosis. Subjects must have pulse oximetry >88% on room air at rest, and a DLco of >49% if there is no evidence of lung metastasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | at least 60 days, and up to 6 months
  The safety of KHK2866 will be determined by reported adverse events (AEs), changes in physical examinations, vital sign measurements, electrocardiograms (ECGs), clinical laboratory evaluations, and treatment discontinuation due to toxicity.

SECONDARY OUTCOMES:
To determine the Cmax, Tmax, AUC and half life of KHK2866 when administered i.v. as monotherapy | at least 28 days and up to 6 months
  Participants will have serial blood samples taken to determine the PK profile of the study drug.
To evaluate the changes in serum HB-EGf in participants administered KHK2866 | at least 60 days, and up to 6 months
  Participants will have serial blood samples taken to develop the PD profile.
To screen for the development of antibodies against KHK2866 (immunogenicity). | at least 60 days and up to 6 months
  Participants will have serial blood samples to check for the development of anti-KHK2866 antibodies.
To describe any anti-tumor activity observed when KHK2866 is administered i.v. as monotherapy, or in combination with chemotherapy. | at least 60 days and up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A Silver, M.D., Study Director — Kyowa Hakko Kirin Pharma, Inc.
Locations (7):
- United States (7):
  - Arizona Cancer Center, Tucson, Arizona
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedar Sinai-Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Oncology Consultants, Houston, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas

REFERENCES:
- [Derived] Sarantopoulos J, Mita MM, Birrer MJ, Cranmer LD, Campos LT, Zhang X, Bristow P, Kaito H, Strout V, Camacho LH. Phase 1 Study of Monotherapy with KHK2866, an Anti-Heparin-Binding Epidermal Growth Factor-Like Growth Factor Monoclonal Antibody, in Patients with Advanced Cancer. Target Oncol. 2016 Jun;11(3):317-27. doi: 10.1007/s11523-015-0394-5. PMID 26507836